CLINICAL TRIAL: NCT03412513
Title: Mirabegron for Treatment of Overactive Bladder Symptoms in Patients With Parkinson's Disease: a Double-blind, Randomized Placebo-controlled Trial
Brief Title: Mirabegron for Treatment of Overactive Bladder Symptoms in Patients With Parkinson's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seung-June Oh, Professor, Department of Urology, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PaDOMi Study
Record Dates: First submitted 2018-01-21; First posted 2018-01-26 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Overactive Bladder; Parkinson Disease
Keywords: Overactive Bladder; Parkinson Disease
MeSH Terms: conditions — Urinary Bladder, Overactive; Parkinson Disease | interventions — mirabegron; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirabegron (Active Comparator): 1:1 randomization to receive Mirabegron 50mg daily or placebo at visit 2. At visit 4 all subjects will receive Mirabegron 50mg.
  Interventions: Drug: Mirabegron
- Placebo (Placebo Comparator): 1:1 randomization to receive Mirabegron 50mg daily or placebo at visit 2. At visit 4 all subjects will receive Mirabegron 50mg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirabegron — Mirabegron 50mg po daily for 12 weeks to Active Comparator group, and 4 weeks(from visit 4 to visit 5) to Placebo comparator group.
  Other Names: Betmiga PR 50mg
  Arms: Mirabegron
Drug: Placebo — Placebo po daily for 8 weeks to Placebo comparator group.
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to see the study drug, Mirabegron, is safe and effective in treating symptoms of Overactive Bladder in patients with Parkinson's disease.

DETAILED DESCRIPTION:
This study is a randomized 1:1 placebo-controlled 12-week study of Mirabegron in 144 Parkinson's subjects the age of 40 to 80 with overactive bladder. Active drug will be Mirabegron 50mg daily. Subjects will be enrolled based on response to an overactive bladder questionnaire at visit 1. Enrolled subjects will have 3 study visits to the clinic as well as 1 phone visit.

ELIGIBILITY:
Inclusion Criteria:

* Subject who signed a consent form approved from IRB(Institutional Review Board) or IEC(Independent Ethics Committee)
* Diagnosis of Parkinson's disease by a neurologist
* taking a Parkinson's medications stably during 4 weeks preceding screening
* 40 Years to 80 Years, Male and Female
* Patient has overactive bladder symptoms more than 4 weeks preceding screening.
* OABSS questionnaires total score≥ 3 and entries of urinary urgency score≥ 2
* The expanded disability status scale ≤ 7

Exclusion Criteria:

* Subjects who have any intervention and operation which can influence on study such as bladder augmentation, vesical sphincter, artificial sphincter, intravesical botulinum toxin treatment etc.
* Use of indwelling catheter or self-catheterization
* acute urinary tract infection or urolithiasis at screening
* History of chronic inflammation such as interstitial cystitis, bladder stones, previous pelvic radiation therapy, or previous or current malignant disease of the pelvic organs
* total volume urine > 3L a day
* Screening post-void residual > 200ml
* Nonpharmacological therapy within the previous 4 weeks of screening
* screening blood pressure >180 systolic or 110 diastolic
* subjects who have orthostatic hypotension, syncope, hypokalemia, or angle-closure glaucoma
* Clinically Significant ECG in recent year
* Screening estimated glomerular filtration rate (eGFR) < 29, AST ( aspartate aminotransferase ) or ALT ( alanine aminotransferase ) > 2x upper limit of normal, γ-GT(gamma-glutamyl transferase) > 3xULN
* take following medication additionally or change the dose: previous 4weeks of screening to end of the study (tamsulosin/silodosin/terazosin, baclofen, diazepam, amitriptyline, DDAVP/desmopressin) previous 12weeks of screening to end of the study (finasteride, dutasteride)
* Use β2- adrenoreceptor agonist, loop diuretic, CYP 3A4 inducer, CYP 2D6 narrow therapeutic index, CYP 3A4 inhibitor, antifungal agent, antiarrhythmic agent
* History of allergy to Mirabegron and beta-adrenergic receptor
* Use of one of the anti-cholinergic bladder medications such as Propiverine / tolterodine / trospium / darifenacin / solifenacin / fesoterodine and mirabegron within 14 days of the screening visit. Subjects who have used one of these medications in the past but discontinued it at least 14 days prior to the screening visit can be enrolled.
* women who have potential to become pregnant during the course of the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-07-16 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the total score of Overactive Bladder Symptom Scale(OABSS) | Baseline(Visit 2 : 0 week), Visit 3(3-5 weeks post Visit 2), Visit 4(6-10 weeks post Visit 2), Visit 5(10-14 weeks post Visit 2)
  Change in the total score of Overactive Bladder Symptom Scale(OABSS) from baseline(Visit 2) to Visit 4

SECONDARY OUTCOMES:
Change in the total score of OABSS(Overactive Bladder Symptom Scale) | Baseline(Visit 2 : 0 week), Visit 3(3-5 weeks post Visit 2), Visit 4(6-10 weeks post Visit 2), Visit 5(10-14 weeks post Visit 2)
  Change in the total score of OABSS, Visit 3, Visit 4 and Visit 5
Change in the total score of IPSS(International Prostate Symptom Score) | Baseline(Visit 2 : 0 week), Visit 3(3-5 weeks post Visit 2), Visit 4(6-10 weeks post Visit 2), Visit 5(10-14 weeks post Visit 2)
  Change in the total score of IPSS and bothersome score, Visit 3, Visit 4 and Visit 5
Change in the total score of OAB-q short form | Baseline(Visit 2 : 0 week), Visit 3(3-5 weeks post Visit 2), Visit 4(6-10 weeks post Visit 2), Visit 5(10-14 weeks post Visit 2)
  Change in the total score of OAB-q short form,Visit 3, Visit 4 and Visit 5
Change in the total score of PPBC(Patient Perception of Bladder Condition) | Baseline(Visit 2 : 0 week), Visit 3(3-5 weeks post Visit 2), Visit 4(6-10 weeks post Visit 2), Visit 5(10-14 weeks post Visit 2)
  Change in the total score of PPBC, Visit 3, Visit 4 and Visit 5
Change in the total score of TSQ (Treatment Satisfaction Questionnaire) | Baseline(Visit 2 : 0 week), Visit 3(3-5 weeks post Visit 2), Visit 4(6-10 weeks post Visit 2), Visit 5(10-14 weeks post Visit 2)
  Change in the total score of TSQ, Visit 3, Visit 4 and Visit 5
Change in the total score of GRA (Global Response Assessment) | Baseline(Visit 2 : 0 week), Visit 3(3-5 weeks post Visit 2), Visit 4(6-10 weeks post Visit 2), Visit 5(10-14 weeks post Visit 2)
  Change in the total score of GRA, Visit 3, Visit 4 and Visit 5
Change in the score of BSW (Benefit, Satisfaction and Willingness to Continue Questions) | Baseline(Visit 2 : 0 week), Visit 3(3-5 weeks post Visit 2), Visit 4(6-10 weeks post Visit 2), Visit 5(10-14 weeks post Visit 2)
  Change in the score of BSW, Visit 4 and Visit 5
Change in the Mean Frequent Urination | Baseline(Visit 2 : 0 week), Visit 3(3-5 weeks post Visit 2), Visit 4(6-10 weeks post Visit 2), Visit 5(10-14 weeks post Visit 2)
  Change in the Mean Frequent Urination, Visit 3 and Visit 4
Change in the Mean number of Urinary urgency | Baseline(Visit 2 : 0 week), Visit 3(3-5 weeks post Visit 2), Visit 4(6-10 weeks post Visit 2), Visit 5(10-14 weeks post Visit 2)
  Change in the Mean number of Urinary urgency, Visit 3 and Visit 4
Change in the Mean number of Urinary incontinence | Baseline(Visit 2 : 0 week), Visit 3(3-5 weeks post Visit 2), Visit 4(6-10 weeks post Visit 2), Visit 5(10-14 weeks post Visit 2)
  Change in the Mean number of Urinary incontinence, Visit 3 and Visit 4

CONTACTS AND LOCATIONS:
Overall Officials: Seung-June Oh, MD, Principal Investigator — Seoul National University Hospital
Locations (5):
- South Korea (5):
  - Kyungpook National University Hospital, Daegu
  - Hallym University Medical Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Severance Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul